CLINICAL TRIAL: NCT04728802
Title: Proxalutamide Treatment for Hospitalized COVID-19 Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KP-DRUG-SARS-003
Record Dates: First submitted 2021-01-27; First posted 2021-01-28 (Actual); Results first posted 2021-06-23 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome)
Keywords: Proxalutamide; Androgen; Anti-androgen
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — proxalutamide

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study.
Who Masked: Participant, Care Provider
Masking Description: Double (Participant, Care Provider)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proxalutamide + Usual Care (Active Comparator): Proxalutamide + usual care as determined by care provider
  Interventions: Drug: Proxalutamide
- Placebo + Usual Care (Placebo Comparator): Placebo + usual care as determined by care provider
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Proxalutamide — Proxalutamide 300mg q.d
  Arms: Proxalutamide + Usual Care
Drug: Placebo — Placebo pill
  Arms: Placebo + Usual Care

SUMMARY:
The purpose of this study is to assess the efficacy and safety of Proxalutamide as a treatment for hospitalized COVID-19 male and female patients.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital with symptoms of COVID-19
2. Male and females age ≥18 years old
3. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization
4. Clinical status on the COVID-19 Ordinal Scale (defined in Section 5.1) of 3, 4, 5, or 6
5. Coagulation: INR ≤ 1.5×ULN, and APTT ≤ 1.5×ULN
6. Subject (or legally authorized representative) gives written informed consent prior to performing any study procedures
7. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

Exclusion Criteria:

1. Subject enrolled in a study to investigate a treatment for COVID-19
2. Requires mechanical ventilation
3. Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc…
4. Patients who are allergic to the investigational product or similar drugs (or any excipients);
5. Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
6. Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
7. Subjects with uncontrolled medical conditions that could compromise participation in the study(e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
8. Known diagnosis of human immunodeficiency virus(HIV) , hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory）
9. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
10. Estimated glomerular filtration rate (eGFR) < 30 ml/min
11. Severe kidney disease requiring dialysis
12. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception, as shown below, throughout the study and for 3 months after stopping GT0918 treatment. Highly effective contraception methods include:

    * Total Abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception, or
    * Use of one of the following combinations (a+b or a+c or b+c):

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS) ;
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository ;
    * Female sterilization (have had prior surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment ;
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient;
    * In case of use of oral contraception women should have been stable for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment, is she considered not of child bearing potential;
13. Sexually active males must use a condom during intercourse while taking the drug and for 3 months after stopping GT0918 treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
14. Subject likely to transfer to another hospital within the next 28 days
15. Subject (or legally authorized representative) not willing or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Cadegiani, MD, Principal Investigator — Applied Biology, Inc.; Andy Goren, MD, Study Director — Applied Biology, Inc.
Locations (8):
- Brazil (8):
  - Hospital Regional José Mendes, Itacoatiara, Amazonas
  - Hospital de Campanha de Manacapuru, Manacapuru, Amazonas
  - Hospital Oscar Nicolau, Manaus, Amazonas
  - Hospital Prontocord, Manaus, Amazonas
  - Hospital Samel, Manaus, Amazonas
  - Hospital Regional Dr. Hamilton Maia Cidae, Manicoré, Amazonas
  - Hospital Raimunda Francisca Dinelli da Silva, Maués, Amazonas
  - Hospital Regional Jofre Cohen, Parintins, Amazonas

IPD SHARING:
Plan to Share IPD: Yes
Yes, study data sets will be made available upon request after peer review and publication.
Supporting Information: Study Protocol, SAP
Time Frame: Available upon request after peer review and publication.
Access Criteria: Available upon request at data@appliedbiology.com

REFERENCES:
- [Background] Goren A, McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Dhurat R, Washenik K, Lotti T. What does androgenetic alopecia have to do with COVID-19? An insight into a potential new therapy. Dermatol Ther. 2020 Jul;33(4):e13365. doi: 10.1111/dth.13365. Epub 2020 Apr 8. No abstract available. PMID 32237190
- [Background] Goren A, Vano-Galvan S, Wambier CG, McCoy J, Gomez-Zubiaur A, Moreno-Arrones OM, Shapiro J, Sinclair RD, Gold MH, Kovacevic M, Mesinkovska NA, Goldust M, Washenik K. A preliminary observation: Male pattern hair loss among hospitalized COVID-19 patients in Spain - A potential clue to the role of androgens in COVID-19 severity. J Cosmet Dermatol. 2020 Jul;19(7):1545-1547. doi: 10.1111/jocd.13443. Epub 2020 Apr 23. PMID 32301221
- [Background] Wambier CG, Vano-Galvan S, McCoy J, Gomez-Zubiaur A, Herrera S, Hermosa-Gelbard A, Moreno-Arrones OM, Jimenez-Gomez N, Gonzalez-Cantero A, Fonda-Pascual P, Segurado-Miravalles G, Shapiro J, Perez-Garcia B, Goren A. Androgenetic alopecia present in the majority of patients hospitalized with COVID-19: The "Gabrin sign". J Am Acad Dermatol. 2020 Aug;83(2):680-682. doi: 10.1016/j.jaad.2020.05.079. Epub 2020 May 22. PMID 32446821
- [Background] Montopoli M, Zumerle S, Vettor R, Rugge M, Zorzi M, Catapano CV, Carbone GM, Cavalli A, Pagano F, Ragazzi E, Prayer-Galetti T, Alimonti A. Androgen-deprivation therapies for prostate cancer and risk of infection by SARS-CoV-2: a population-based study (N = 4532). Ann Oncol. 2020 Aug;31(8):1040-1045. doi: 10.1016/j.annonc.2020.04.479. Epub 2020 May 6. PMID 32387456
- [Background] McCoy J, Cadegiani FA, Wambier CG, Herrera S, Vano-Galvan S, Mesinkovska NA, Ramos PM, Shapiro J, Sinclair R, Tosti A, Goren A. 5-alpha-reductase inhibitors are associated with reduced frequency of COVID-19 symptoms in males with androgenetic alopecia. J Eur Acad Dermatol Venereol. 2021 Apr;35(4):e243-e246. doi: 10.1111/jdv.17021. Epub 2020 Nov 22. No abstract available. PMID 33135263
- [Background] McCoy J, Wambier CG, Herrera S, Vano-Galvan S, Gioia F, Comeche B, Ron R, Serrano-Villar S, Iwasiow RM, Tayeb MA, Cadegiani FA, Mesinkovska NA, Shapiro J, Sinclair R, Goren A. Androgen receptor genetic variant predicts COVID-19 disease severity: a prospective longitudinal study of hospitalized COVID-19 male patients. J Eur Acad Dermatol Venereol. 2021 Jan;35(1):e15-e17. doi: 10.1111/jdv.16956. Epub 2020 Oct 21. No abstract available. PMID 32977355
- See also: The AndroCoV Project — http://appliedbiology.com/AppliedBiologyTheAndroCoVProject.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
Started | 317 | 328
Completed (All randomized patients were included in analysis) | 288 | 292
Not Completed | 29 | 36
Not completed — Withdrawal by Subject | 4 | 20
Not completed — Physician Decision | 7 | 7
Not completed — Protocol Violation | 10 | 4
Not completed — Transfer | 1 | 0
Not completed — Death | 4 | 5
Not completed — Other | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care | Total
Number analyzed (Participants) | 317 | 328 | 645
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 50 [41 to 62] | 49 [38 to 61] | 50 [39 to 61.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 133 | 146 | 279
  Male | 184 | 182 | 366
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 317 | 328 | 645
Body mass index over 30 kg/m2 [Count of Participants; unit: Participants] | 28 | 25 | 53
Hypertension [Count of Participants; unit: Participants] | 93 | 82 | 175
Type 2 diabetes mellitus [Count of Participants; unit: Participants] | 41 | 38 | 79
Chronic obstructive pulmonary disorder [Count of Participants; unit: Participants] | 8 | 8 | 16
Chronic kidney disease [Count of Participants; unit: Participants] | 0 | 0 | 0
0 Coexisting conditions [Count of Participants; unit: Participants] | 204 | 227 | 431
1 Coexisting conditions [Count of Participants; unit: Participants] | 68 | 56 | 124
2+ Coexisting conditions [Count of Participants; unit: Participants] | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: 14 Day Recovery Rate
Description: Recovery rate defined as those reaching scores 1 or 2 over 14 days after randomization on the COVID-19 ordinal scale.
  The ordinal scale is defined as follows:
  8. Death; 7. Hospitalized, on invasive mechanical ventilation or ECMO; 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5. Hospitalized, requiring supplemental oxygen; 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise; 3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2. Not hospitalized, limitation on activities;
  1. Not hospitalized, no limitations on activities
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 317 | 328
Participants | 258 | 117

2. Secondary Outcome: 28 Day Recovery Rate
Description: Recovery rate defined as those reaching scores 1 or 2 over 28 days after randomization on the COVID-19 ordinal scale.
  The ordinal scale is defined as follows:
  8. Death; 7. Hospitalized, on invasive mechanical ventilation or ECMO; 6. Hospitalized, on non-invasive ventilation or high flow oxygen devices; 5. Hospitalized, requiring supplemental oxygen; 4. Hospitalized, not requiring supplemental oxygen- requiring ongoing medical care (COVID-19 related or otherwise; 3. Hospitalized, not requiring supplemental oxygen - no longer requires ongoing medical care; 2. Not hospitalized, limitation on activities;
  1. Not hospitalized, no limitations on activities
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 317 | 328
Participants | 271 | 155

3. Secondary Outcome: 28 Day Mortality Rate
Description: All-cause mortality rate over 28 days post randomization.
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 317 | 328
Participants | 35 | 162

4. Secondary Outcome: Post-Randomization Time to Recover (Alive Hospital Discharge)
Description: Number of day post-randomization required to achieve live hospital discharge.
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
Number analyzed (Participants) | 317 | 328
Days | 5 [3 to 8] | 10 [6 to 15]

ADVERSE EVENTS:
Time Frame: 28 Days
Arm/Group | Proxalutamide + Usual Care | Placebo + Usual Care
All-Cause Mortality (participants affected / at risk) | 35/317 | 162/328
Serious Adverse Events (participants affected / at risk) | 38/317 | 170/328
Other Adverse Events (participants affected / at risk) | 51/317 | 11/328
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Proxalutamide + Usual Care (N=317) | Placebo + Usual Care (N=328)
Death (General disorders) | 35 | 162
Mechanical Ventilation (Respiratory, thoracic and mediastinal disorders) | 5 | 41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Proxalutamide + Usual Care (N=317) | Placebo + Usual Care (N=328)
Diarrhea (Gastrointestinal disorders) | 51 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT04728802/Prot_SAP_001.pdf